CLINICAL TRIAL: NCT01451515
Title: NHL16: Study For Newly Diagnosed Patients With Acute Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL16; NCI-2012-00496 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2011-08-17; First posted 2011-10-13 (Estimated); Results first posted 2022-05-23 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Lymphoblastic Lymphoma
Keywords: Lymphoblastic lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Prednisolone; Vincristine; Daunorubicin; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Doxorubicin; Cyclophosphamide; Cytarabine; Thioguanine; Clofarabine; Methotrexate; Mercaptopurine; Dexamethasone; Calcium Dobesilate; Hydrocortisone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will undergo treatment as described in the intervention section. Interventions include:
  * Remission induction: prednisone, vincristine, daunorubicin, PEG-asparaginase (or Erwinia asparaginase), IT-MHA (Methotrexate, hydrocortisone, and cytarabine), cyclophosphamide, cytarabine, thioguanine
  * Consolidation: PEG-asparaginase, High-dose methotrexate (HD-MTX), mercaptopurine
  * Postremission continuation: Dexamethasone, doxorubicin, vincristine, mercaptopurine, PEG-asparaginase, cyclophosphamide, cytarabine, methotrexate
  * Reintensification: dexamethasone, cytarabine, etoposide, PEG-asparaginase, clofarabine, cyclophosphamide
  * All patients receive IT-MHA on days 1 and 15. Some patients also receive additional IT-MHA on days 8 and 22.
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Daunorubicin; Drug: PEG-asparaginase; Drug: Erwinia asparaginase; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Thioguanine; Drug: Clofarabine; Drug: Methotrexate; Drug: Mercaptopurine; Drug: Dexamethasone; Drug: Hydrocortisone; Drug: Etoposide

INTERVENTIONS:
Drug: Prednisone — Given orally (PO).
  Other Names: Prednisolone
Drug: Vincristine — Given intravenously (IV).
  Other Names: Oncovin®; Vincristine sulfate
Drug: Daunorubicin — Given IV.
  Other Names: Daunomycin; Cerubidine®
Drug: PEG-asparaginase — Given intramuscularly (IM) or IV.
  Other Names: Pegaspargase; Oncaspar®
Drug: Erwinia asparaginase — Given IM or IV if allergy occurs with the first or second PEG-asparaginase dose.
  Other Names: Erwinase®
Drug: Doxorubicin — Given IV.
  Other Names: Adriamycin®
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
Drug: Cytarabine — Given IV or IT.
  Other Names: Ara-C; Cytosar-U®
Drug: Thioguanine — Given PO.
  Other Names: Purine antimetabolite
Drug: Clofarabine — Given IV.
  Other Names: Cl-F-Ara-A; CAFdA; 2-Chloro-9-(2-deoxy-2-fluoro-beta-D-arabinofuranosyl)-9H-purin-6-amine; Clofarex; Clolar^TM
Drug: Methotrexate — Given IV, IM or IT.
  Other Names: MTX; High-dose methotrexate (HD-MTX)
Drug: Mercaptopurine — Given PO.
  Other Names: 6-MP; Purinethol®
Drug: Dexamethasone — Given PO or IV.
  Other Names: Decadron®
Drug: Hydrocortisone — Given IT.
  Other Names: Cortef®
Drug: Etoposide — Given IV.
  Other Names: VP-16; Vepesid®

SUMMARY:
This is a phase II clinical trial using risk-adapted therapy. The treatment is acute lymphoblastic leukemia (ALL)-based therapy, using multi-agent regimens comprising of induction, consolidation, and continuation (maintenance) phases delivered over 24-30 months. Participants will be classified into 3 treatment stratums, based on bone marrow/peripheral blood lymphoma cells involvement at diagnosis and day 8 for T-lymphoblastic lymphoma and bone marrow/peripheral blood lymphoma cells involvement at diagnosis for B-lymphoblastic lymphoma.

The Primary Objective of this study is:

To improve the outcome of children with lymphoblastic lymphoma (LL) who have minimal disseminated disease (MDD) equal to or more than 1% at diagnosis by using MDD- and minimal residual disease (MRD)- based risk-adapted therapy.

The Secondary Objectives of this study are:

* To estimate the event-free survival and overall survival of children with lymphoblastic lymphoma who are treated with MDD- or MRD-based risk- directed therapy.
* To evaluate the prognostic value of levels of MDD at diagnosis and MRD on day 8 of remission induction.

DETAILED DESCRIPTION:
TREATMENT PLAN

Treatment will consist of 3 main phases: remission induction, consolidation [only for patients with any central nervous system (CNS) disease and/or testicular involvement], and continuation.

* Induction (6-7 weeks).
* Consolidation for participants with CNS involvement or those with testicular disease only (10 weeks).
* Reintensification - Participants with residual disease any time after induction therapy may receive 1-2 cycles of re-intensification therapy and may proceed to allogeneic stem cell transplant if suitable donor is available.
* Continuation Therapy (98-120 weeks).
* Intrathecal Chemotherapy (days 1 and 15; if needed also on days 8 and 22)

TREATMENT SCHEME

T lymphoblastic lymphoma: bone marrow/peripheral blood (BM/PB) involvement (MDD/MRD): Diagnosis: less than 1%; Day 8: +/- (Stratum 1)

* Induction

  * Single dose of Cyclophosphamide
  * Steroid: prednisone
* Continuation: 98 weeks

T lymphoblastic lymphoma: BM/PB involvement (MDD/MRD): Diagnosis: equal to or greater than 1%; Day 8: - (Stratum 2)

* Induction

  * Fractionated Cyclophosphamide
  * Steroid: prednisone
* Continuation : 98 weeks

T lymphoblastic lymphoma: BM/PB involvement (MDD/MRD): Diagnosis: equal to or greater than 1%; Day 8: + (Stratum 3)

* Induction

  * Fractionated Cyclophosphamide
  * Steroid: prednisone and dexamethasone
* Continuation: 120 weeks

B lymphoblastic lymphoma: Stage I-III (Stratum 1)

* Induction

  * Single dose of Cyclophosphamide
  * Steroid: prednisone
* Continuation: 98 weeks

B lymphoblastic lymphoma: Stage IV or testicular (Stratum 2)

* Induction

  * Fractionated Cyclophosphamide
  * Steroid: prednisone
* Continuation: 98 weeks

Patients with CNS or testicular involvement will receive Consolidation therapy prior to continuation therapy and receive extended maintenance therapy (120 weeks).

Any patient with detectable disease (MRD, bone marrow or biopsy of residual mass) at the end of induction may be considered for reintensification and/or hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of newly diagnosed lymphoblastic lymphoma (patients must have <25% tumor cells in bone marrow by morphology)
2. Age ≤ 21 years
3. Limited prior therapy, including systemic glucocorticoids for 1 week or less, 1 dose of vincristine, emergency radiation therapy to the mediastinum, and 1 dose of IT chemotherapy. Other circumstances must be cleared by PI or co-PI.
4. Written, informed consent and assent following guidelines of the Institutional Review Board, National Cancer Institute (NCI), Food and Drug Administration (FDA), and Office of Human Research Protections (OHRP).

Exclusion Criteria:

1. Participants with prior therapy, other than therapy specified in 3 above.
2. Participants who are pregnant or lactating.
3. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroto Inaba, MD,PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Rady Children's Hospital San Diego, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 eligible patients were recruited between 23MAY2012 and 06DEC2016
Groups:
- Stratum 1: Minimal disseminated disease (MDD) <1% at diagnosis in T-lymphoblastic lymphoma No bone marrow involvement microscopically at diagnosis in B-lymphoblastic lymphoma
  Patients should not have:
  * Any CNS involvement: CNS-3 status (i.e., ≥5 WBC/µL of CSF with blasts or cranial nerve palsy), CNS-2 status (<5 WBC/µL of CSF with blasts) or traumatic LP (>10 RBC/µL of CSF with blasts)
  * Overt testicular involvement (evidenced by ultrasonogram).
- Stratum 2: * MDD ≥1% and MRD negative (<0.01%) on day 8 in T-lymphoblastic lymphoma
  * Bone marrow involvement microscopically present at diagnosis in B-lymphoblastic lymphoma
  * Any CNS involvement: CNS-3 status (i.e., ≥5 WBC/µL of CSF with blasts or cranial nerve palsy), CNS-2 status (<5 WBC/µL of CSF with blasts) or traumatic LP (>10 RBC/µL of CSF with blasts) but does not fulfill the criteria of stratum 3
  * Overt testicular involvement (evidenced by ultrasonogram) but does not fulfill the criteria of stratum 3
- Stratum 3: Any patients with MDD ≥1% and MRD positive (≥0.01%) on day 8 in T-lymphoblastic lymphoma
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Started | 12 | 7 | 4
Completed | 11 | 4 | 3
Not Completed | 1 | 3 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Development of unacceptable toxicity during treatment | 0 | 0 | 1
Not completed — Relapse (except CNS) | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3 | Total
Number analyzed (Participants) | 12 | 7 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.23 (4.48) | 11.27 (5.73) | 12.58 (4.43) | 12.00 (4.69)
Age, Continuous [Median (Full Range); unit: years] | 13.0 [4.50 to 17.95] | 12.3 [3.66 to 19.63] | 13.0 [6.75 to 17.52] | 12.9 [3.66 to 19.63]
Age, Customized [Count of Participants; unit: Participants]
  <10 years | 5 | 2 | 1 | 8
  >=10 years | 7 | 5 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 9
  Male | 7 | 4 | 3 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 4 | 3 | 17
  Black | 2 | 2 | 1 | 5
  Multiple Race (NOS) | 0 | 1 | 0 | 1
  NOS Spanish,Hispanic,Latino | 0 | 1 | 0 | 1
  Non Spanish speaking, Non Hispanic | 12 | 6 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Probability of Event-free Survival (EFS)
Description: For EFS, relapse and second malignancies are considered as failures in addition to death in complete remission. The time to EFS will be set to 0 for patients who fail to achieve complete remission. Kaplan-Meier estimates of the OS and EFS curves are computed, along with estimates of standard errors by Peto's method.
  Please note the unit of measurement of probabilities are percentages.
Time Frame: Two years post therapy.
Measure: Number (95% Confidence Interval); unit: percentage of event-free patients
Groups:
- All Enrollments: Twenty-three (23) eligible patients
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3 | All Enrollments
Number analyzed (Participants) | 12 | 7 | 4 | 23
percentage of event-free patients | 91.7 [53.9 to 98.8] | 71.4 [25.8 to 92.0] | 100 [100 to 100] | 86.96 [64.81 to 95.60]

2. Secondary Outcome: Probability of Overall Survival (OS)
Description: For OS, only deaths are considered failures for OS. Kaplan-Meier estimates of the OS curves are computed along with estimates of standard errors by Peto's method.
  Please note the unit of measurement of probabilities are percentages.
Time Frame: Two years post therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3 | All Enrollments
Number analyzed (Participants) | 12 | 7 | 4 | 23
percentage of patients alive | 91.7 [53.9 to 98.8] | 71.4 [25.8 to 92.0] | 100 [100 to 100] | 86.96 [64.81 to 95.60]

3. Secondary Outcome: Minimal Disseminated Disease (MDD)
Description: Detectable disease in bone marrow or blood: A binary measure, positive (detectable), negative (non-detectable)
Time Frame: At Diagnosis
Population: Fourteen patients had MDD data at diagnosis.
Measure: Number; unit: participants
Groups:
- Stratum 2: MDD ≥1% and MRD negative (<0.01%) on day 8 in T-lymphoblastic lymphoma
  * Bone marrow involvement microscopically present at diagnosis in B-lymphoblastic lymphoma
  * Any CNS involvement: CNS-3 status (i.e., ≥5 WBC/µL of CSF with blasts or cranial nerve palsy), CNS-2 status (<5 WBC/µL of CSF with blasts) or traumatic LP (>10 RBC/µL of CSF with blasts) but does not fulfill the criteria of stratum 3
  * Overt testicular involvement (evidenced by ultrasonogram) but does not fulfill the criteria of stratum 3
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Number analyzed (Participants) | 5 | 5 | 4
participants
  Negative | 4 | 2 | 0
  Positive | 1 | 3 | 4

4. Secondary Outcome: Minimal Residual Disease (MRD)
Description: Detectable disease in bone marrow or blood: A binary measure, positive (detectable), negative (non-detectable)
Time Frame: Day 8
Population: Seventeen participants had MRD data at day 8
Measure: Number; unit: participants
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Number analyzed (Participants) | 8 | 5 | 4
participants
  Negative | 8 | 4 | 0
  Positive | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: From the start of treatment to 30 days after the last treatment is taken. Treatment last for 2 to 2½ years.
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3 | All Enrollments
All-Cause Mortality (participants affected / at risk) | 2/12 | 2/7 | 0/4 | 4/23
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/7 | 0/4 | 1/23
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7 | 4/4 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=12) | Stratum 2 (N=7) | Stratum 3 (N=4) | All Enrollments (N=23)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 (N=12) | Stratum 2 (N=7) | Stratum 3 (N=4) | All Enrollments (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 4 | 4 | 19
Upper respiratory infection (Infections and infestations) | 10 | 3 | 3 | 16
Mucosal Infection (Infections and infestations) | 5 | 2 | 1 | 8
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 8 | 4 | 3 | 15
Skin infection (Infections and infestations) | 6 | 3 | 1 | 10
Alanine aminotransferase increased (Investigations) | 4 | 2 | 1 | 7
Fever (General disorders) | 5 | 3 | 1 | 9
Blood bilirubin increased (Investigations) | 4 | 1 | 1 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 8
Sinusitis (Infections and infestations) | 5 | 2 | 1 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0 | 2 | 7
Otitis media (Infections and infestations) | 4 | 2 | 1 | 7
Lipase increased (Investigations) | 1 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 6
Depression (Psychiatric disorders) | 2 | 2 | 3 | 7
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 5
Cholesterol high (Investigations) | 2 | 1 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 0 | 6
Neuralgia (Nervous system disorders) | 3 | 4 | 1 | 8
Hypotension (Vascular disorders) | 3 | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Enterocolitis infectious (Infections and infestations) | 1 | 2 | 2 | 5
Lung infection (Infections and infestations) | 3 | 1 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 6
Colitis (Gastrointestinal disorders) | 2 | 2 | 2 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 5
Serum amylase increased (Investigations) | 1 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2 | 0 | 3
Paronychia (Infections and infestations) | 2 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 2
Pain (General disorders) | 2 | 0 | 1 | 3
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 0 | 1 | 3
Wound infection (Infections and infestations) | 0 | 2 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 1 | 3
Syncope (Nervous system disorders) | 2 | 1 | 0 | 3
Thromboembolic event (Vascular disorders) | 1 | 1 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Rectal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Allergic reaction (Immune system disorders) | 1 | 1 | 0 | 2
Allergic reaction to Asparaginase (Immune system disorders) | 1 | 0 | 1 | 2
Lip infection (Infections and infestations) | 1 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
GGT increased (Investigations) | 2 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 1 | 2
Seizure (Nervous system disorders) | 1 | 1 | 0 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0 | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Edema limbs (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Anaphylaxis (Immune system disorders) | 0 | 0 | 1 | 1
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Small intestine infection (Infections and infestations) | 1 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Radiculitis (Nervous system disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT01451515/Prot_SAP_000.pdf